CLINICAL TRIAL: NCT03155542
Title: Alcohol Intake, Alcohol Metabolizing Enzymes Gene Polymorphisms and the Risk of Colorectal Cancer
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 201610059RIND
Record Dates: First submitted 2017-05-14; First posted 2017-05-16 (Actual); Last update posted 2017-05-23 (Actual); Status verified 2017-05

CONDITIONS: Colorectal Neoplasms
Keywords: alcohol; gene polymorphisms; Colorectal cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — 5-10 ml venous blood sample
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- colorectal cancer patient case group: Histologically confirmed colorectal adenocarcinoma
- family member control group: without the diagnosis of CRC and accompanied the patient to the primary care clinic visit

SUMMARY:
According to the statistic reports from World Health Organization (WHO) International Agency for Research on Cancer (IARC), the incidence and mortality rate of colorectal cancer ranked third and fourth respectively among ten most commonly diagnosed cancer worldwide; moreover, based on the statistics from Health Promotion Administration, Ministry of Health and Welfare in Taiwan, the incidence and mortality rate of colorectal cancer ranked second and third respectively among call cancer in Taiwanese population. However, if colorectal cancer is diagnosed and treated in early phase, the 5-year survival rate for stage I colorectal cancer can be up to 90%; on the other hand, the 5-year survival rate for end stage colorectal cancer is only approximately 10%. Therefore, the screening, early diagnosis od colorectal cancer is crucial. To date, there are some known risk factors for colorectal cancer, including familial adenomatous polyposis, obesity, physical inactivity, etc. Alcohol had also been identified as an important risk factor for colorectal cancer, and the risk could be higher among Asian population because of the reduced enzymatic activity of some of the alcohol metabolizing enzymes. Thus, through this study, the investigators hope to find out the risk factors of colorectal cancer among Taiwanese population, including alcohol metabolizing enzyme gene polymorphisms and their interaction with environmental factors, to attain the purpose of early prevention of colorectal cancer.

DETAILED DESCRIPTION:
The purpose of this study is to find out relationship between alcohol metabolizing enzyme gene polymorphism and colorectal cancer, and discuss the impact of the interaction between gene polymorphism and environmental factors on the risk of colorectal cancer.

ELIGIBILITY:
Inclusion criteria:

Case:

* Histologically confirmed colorectal adenocarcinoma at National Taiwan University Hospital (NTUH) from 2000 to 2016
* Age >20 at the time of inclusion

Control:

* No diagnosis of colorectal cancer
* Age >20 at the time of inclusion
* Family members of case, including parents, siblings, offspring, spouse mother-in-law or daughter-in-law

Exclusion criteria (Both for case and control):

* History of familial adenomatous polyposis
* History of partial or total removal of the colorectum
* History of inflammatory bowl disease
* History of malignant neoplasms

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: primary care clinic visit at National Taiwan University Hospital
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-03-22 (Actual); Study Completion 2017-03-29 (Actual)

PRIMARY OUTCOMES:
colorectal cancer diagnosis | 4 months
  Histologically confirmed colorectal adenocarcinoma

CONTACTS AND LOCATIONS:
Overall Officials: Yen-Hui CHEN, Principal Investigator — Graduate Institute of Clinical Pharmacy, College of Medicine, National Taiwan University
Locations (1):
- National Taiwan University Hospital, Taipei, ROC, Taiwan

IPD SHARING:
Plan to Share IPD: No